CLINICAL TRIAL: NCT05597995
Title: A Prospective Clinical Trial Evaluating the Efficacy of 1.5% Sodium Tetradecyl Sulfate Foam Injection for the Treatment of Epidermoid Cysts
Brief Title: Treatment of Epidermoid Cysts
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EIC-STS
Record Dates: First submitted 2022-10-20; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Epidermoid Cyst
Keywords: epidermoid; cyst; epidermoid cyst; small bumps beneath skin
MeSH Terms: conditions — Epidermal Cyst; Cysts | interventions — Sodium Tetradecyl Sulfate

STUDY DESIGN:
Intervention Model Description: Enrolled subjects will undergo aspiration of cyst contents through an 18g needle immediately followed by injection of 1.5% STS foam (until the cyst is full and foam is flowing out of the injection site) followed by surgical excision 60 days later. The foam will be created by diluting 3% STS with an equal volume of normal saline then mixing with air in a 1:4 ratio using a female-to-female coupler.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment with 1.5% sodium tetradecyl sulfate foam (Experimental): each subject will have cyst contents aspirated through an 18g needle followed by an injection of 1.5% STS solution foamed 1:4 with air until foam is flowing out of the injection site.
  Interventions: Drug: Sodium Tetradecyl Sulfate

INTERVENTIONS:
Drug: Sodium Tetradecyl Sulfate — subjects epidermoid cysts will be treated with 1.5% sodium tetradecyl sulfate foam
  Other Names: 1.5% sodium tetradecyl sulfate foam

SUMMARY:
The objective of this study is to determine the efficacy, safety, tolerability, and patient satisfaction associated with the treatment of epidermoid cysts with injected 1.5% sodium tetradecyl sulfate (STS) foam.

DETAILED DESCRIPTION:
The primary objective is to determine the efficacy of STS foam injection on EIC with an endpoint of clinical resolution and cyst wall destruction on histology.

Enrolled subjects will undergo aspiration of cyst contents through an 18g needle immediately followed by injection of 1.5% STS foam (until the cyst is full and foam is flowing out of the injection site) followed by surgical excision 60 days later. The foam will be created by diluting 3% STS with an equal volume of normal saline then mixing with air in a 1:4 ratio using a female-to-female coupler.

ELIGIBILITY:
Inclusion Criteria:

* Adults in good general health based on the investigator's judgment and medical history aged 18-80 years old
* Must be willing to sign a photography release and ICF.
* Subject must be willing to undergo study procedures, including STS foam injection and excision with simple closure with an expected linear scar.
* Epidermal inclusion cyst on the skin (not on mucosa or genitals) at least 4 mm in size
* Negative urine pregnancy test at the time of study entry (if applicable)
* Females will be either of non-childbearing potential defined as:

  1. Having no uterus
  2. No menses for at least 12 months. Or; Female subjects of childbearing potential must agree to use an effective method of birth control during the course of the study. All systemic birth control measures must be in consistent use for at least 30 days prior to study enrollment participation. Acceptable forms of birth control are below:

  <!-- -->

  1. Oral contraceptive pill, injection, implant, patch, vaginal ring, intrauterine device
  2. Intrauterine coil
  3. Bilateral tubal ligation
  4. Hysterectomy
  5. Barrier method used with an additional form of contraception (e.g., sponge, spermicide, or condom)
  6. Abstinence (If practicing abstinence, must agree to use a barrier method described above (4) If they become sexually active).
  7. Vasectomized (must agree to use barrier method described above (4) if they become sexually active with an un-vasectomized partner).

Exclusion Criteria:

* Pregnancy or planned pregnancy during the study or currently breastfeeding.
* Previously excised cysts or actively inflamed cysts will not be included in the study.
* Presence of incompletely healed wound in the treatment area.
* Any UNCONTROLLED systemic disease -a potential patient in whom therapy for a systemic disease is not yet stabilized will not be considered for entry into the study.
* Significant history or current evidence of a medical, psychological, or other disorder that, in the investigator's opinion, would preclude enrollment into the study.
* Allergy to STS.
* Active dermatitis, active bacterial, neurologic, fungal, or viral infection in the proposed treatment area.
* Inability to ambulate following the procedure.
* Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Investigator Assessment of EIC (Epidermal inclusion cysts) resolution | Day 60
  Investigator Assessment of EIC (Epidermal inclusion cysts) resolution or recurrence Did the cyst resolve (involution or substantial decrease in size and clinical appearance)?
  (circle one)
  Resolved Did not resolve
Cyst wall destruction on histologic examination as determined by a board-certified dermatopathologist | Day 60
  A dermatopathologist will examine the excised cysts to determine if the cyst lining was damaged by injection of STS foam, as demonstrated by the presence of necrotic squamous epithelium.

SECONDARY OUTCOMES:
Subject satisfaction rating | Day 60
  1. Extremely satisfied
  2. Satisfied
  3. Slightly satisfied
  4. Slight dissatisfied
  5. Dissatisfied
  6. Extremely satisfied
Investigator skin irritation assessment (Draize scale) | Baseline, Day 1, Day 7
  Investigator skin irritation assessment (Draize scale) Score Erythema Edema
  0 No erythema No Edema
  1. Very slight Erythema very slight edema
  2. Well-defined erythema Well-defined Edema
  3. Moderate-to-severe erythema Moderate edema (raised approx 1mm)
  4. Severe erythema (beet redness) Severe edema (raised greater than 1mm and extending beyond area of exposure)
Subject injection site pain assessment on visual analog scale | Baseline, Day 1, Day 7
  Visual Analog Scale
  Rate your pain on a scale of 1 to 10 ( circle one)
  1 2 3 4 5 6 7 8 9 10

IPD SHARING:
Plan to Share IPD: Undecided